CLINICAL TRIAL: NCT06645535
Title: The Role and Mechanism of Gut Microbiota and Metabolites in Heart Failure With Preserved Ejection Fraction
Brief Title: The Gut Microbiota and Metabolites in HFpEF
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Lei Zhou, Director of Geriatric Cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: HFpEF 001
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: gut microbiota; metabolites; HFpEF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum samples, and stool samples were obtained from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF group: Patients with heart failure with preserved ejection fraction.
- HFrEF group: Patients with heart failure with reduced ejection fraction.
- Control group: Control participants without heart failure.

SUMMARY:
Heart failure (HF) with preserved ejection fraction (HFpEF) has emerged as a critical public health concern. The annual mortality rate for HFpEF is approximately 15%, accompanied by a re-hospitalization rate of nearly 80%. Survival rates over a 5-year period typically range from 25% to 50%. Existing medications effective against HF with reduced ejection fraction (HFrEF) have shown no significant effect on HFpEF. Only the sodium-glucose cotransporter 2 inhibitor (SGLT2i) has demonstrated significant improvements in patient survival and re-hospitalization rates, thus earning a Class IA recommendation in clinical guidelines. HFpEF is characterized as a complex, heterogeneous, multi-organ systemic syndrome primarily associated with risk factors such as advanced age, obesity, metabolic syndrome, type 2 diabetes mellitus (T2DM), hypertension, sedentary lifestyle, coronary atrial disease (CAD), and kidney disease. Therefore, it is crucial to investigate other multi-system disorders closely associated with cardiac diastolic dysfunction to gain a comprehensive understanding of the underlying mechanisms of HFpEF. The human digestive tract harbors a complex and dynamic microbial community known as the gut microbiota, which comprises up to 100 trillion microorganisms and approximately 150 times more genomes than the human genome, often referred to as the "second genome" of the human body. Recent years have seen growing recognition and extensive research into the role of gut microbiota in the pathogenesis and development of cardiovascular diseases. In HFrEF patients, there is a significant decrease in the diversity of gut microbiota, along with changes in its composition and structure. Notably, pathogenic bacteria such as Campylobacter and Candida species exhibit a substantial increase correlating with disease severity, while anti-inflammatory bacteria like Brauteria demonstrate a marked decrease. Furthermore, gut microbiota can influence the host's cardiometabolic traits through the modulation of both its own and host-produced metabolites. HFpEF is increasingly considered a metabolic disease. Comorbidities associated with HFpEF, including obesity, T2DM, metabolic syndrome, hypertension, and coronary artery disease (CAD), have been reported to be closely related to gut microbiota. However, the relationship between gut microbiota and HFpEF is still not fully understood. A recent study indicates that indole-3-propionic acid (IPA) could attenuate diastolic and metabolic dysfunction and mitigate gut microbiota dysbiosis in an HFpEF mouse model. Several clinical studies have noted alterations in microbial metabolites such as short-chain fatty acids (SCFAs), and trimethylamine N-oxide (TMAO) in HFpEF patients. It is now well recognized that targeting the gut microbiome and its metabolites represents a promising novel therapeutic strategy for managing cardiovascular diseases. Therefore, this study is to investigate the changes and function of gut microbiota and metabolites in HFpEF.

DETAILED DESCRIPTION:
1. Heart failure with preserved ejection fraction is an urgent clinical challenge As the leading killer of human life and health, cardiovascular disease is a difficult public health problem worldwide. According to the latest statistics of China Cardiovascular Health and Disease Report 2022, the number of patients in China has exceeded 330 million, and the number of patients with heart failure (HF) is as high as 8.9 million, becoming the second leading cause of death related to heart disease after coronary heart disease. According to the 2023 European Society of Cardiology (ESC) guidelines for the diagnosis and management of acute and chronic heart failure, LVEF) classified heart failure into three categories: heart failure with reduced ejection fraction (HFrEF, LVEF≤40%), and heart failure with reduced ejection fraction (HfreF). heart failure with mildly reduced ejection fraction (HFmrEF, Heart failure with mildly reduced ejection fraction) 40% < LVEF < 49%) and heart failure with preserved ejection fraction (HFpEF, EF≥50%). Among them, HFpEF accounts for about 50% of all heart failure, and with the improvement of HFpEF cognition and diagnosis rate, and the aggravation of population aging, its prevalence shows an increasing trend year by year. The annual mortality rate is about 15%, the rehospitalization rate is up to 80% within 5 years after hospitalization, and the survival rate is only 25%-50%. At present, the diagnosis and treatment system of HFrEF is maturing, and the quality of life and overall prognosis of patients are gradually improving. However, there are effective therapeutic drugs for HFrEF. These include angiotensin receptor neprilysin inhibitor (ARNi), angiotensin receptor blocker (angiotensin receptor blocker), and angiotensin receptor inhibitor (ARNI). ARB), Mineralocorticoid Receptor Antagonists (MRAs), PDE-5 inhibitors, etc., have no significant effect on HFpEF. Only one HFpEF positive clinical drug, sodium glucose cotransporter 2 inhibitor (SGLT2i), significantly improved patient survival and rehospitalization rate, and was included in the class IA recommendation of the guidelines. The pathogenesis of HFpEF is complex, and the clinical diagnosis and treatment methods are limited. The incidence and rehospitalization rate of HFpef are increasing year by year, resulting in serious social and economic losses and disease burden. Therefore, exploring the pathogenesis of HFpEF and finding effective prevention and treatment methods are major clinical scientific problems that need to be solved urgently.
2. Clinical characteristics and risk factors of HFpEF HFpEF is not a single heart disease, but a complex, heterogeneous, multi-organ, systemic syndrome. It is often associated with patients with advanced age, obesity, metabolic syndrome, type 2 diabetes, hypertension, sedentary behavior, coronary heart disease, and kidney disease. Among them, hypertension and coronary heart disease are common risk factors for HFrEF and HFpEF, while people with obesity, abnormal metabolism and lack of physical activity are more likely to develop HFpEF. Although studies on HFpEF are increasing, little progress has been made in the treatment of HFpEF. At present, the only drug that has been proven to effectively improve the prognosis of patients is SGLT2i, and the primary indication is for patients with type 2 diabetes, further indicating that metabolic disorders such as diabetes are closely related to HFpEF. Systemic inflammation, metabolic disorders, vascular dysfunction, oxidative stress and other factors induce cardiomyocyte hypertrophy, myocardial fibrosis, and intracellular calcium processing disorders, which lead to myocardial active relaxation dysfunction and cardiomyocyte stiffness, and then the decline of left ventricular diastolic function, abnormal left ventricular filling, decreased myocardial compliance, and cardiac overload leading to HFpEF. The dysfunction and metabolic disorders of HFpEF involve multiple organs outside the heart. Therefore, the study of the mechanism of HFpEF should not be limited to the cardiac level.
3. Gut microbiota is closely related to cardiovascular disease Gut microbiota is a complex and dynamic microbial community inhabiting in the human digestive tract. The total number of microorganisms inhabiting in the human gut is up to 100 trillion, and the total number of genomes is about 150 times that of the human genome, which is called the "second genome" of the human body. According to the existing research data, the gut microbiota is generally divided into six major phyla, namely Firmicutes, Bacteroidetes, Actinobacteria, Proteobacteria, Fusobacteria and Verrucomicrobia. Firmicutes and Bacteroidetes are the main types. The main functions of gut microbiota include: fermentation of incompletely digested food, synthesis of certain vitamins, fermentation of sugars to produce Short Chain Fatty Acids (SCFAs) such as acetic acid, propionic acid and butyric acid, and regulation of intestinal epithelial mucosal barrier and immune system. In the healthy state, various microorganisms maintain symbiotic or antagonistic relationships in the intestinal tract, forming the microbial homeostasis of the human gastrointestinal tract, which plays an important role in the regulation of the host body's metabolism, nutrition, and immunity. Unhealthy diet, drugs and lifestyle can lead to the imbalance of intestinal flora and induce a variety of diseases. Therefore, the balance of intestinal flora is closely related to human diseases and health. In recent years, with the development and application of 16S rDNA sequencing technology, metagenomic sequencing technology and metabolomics, the role of intestinal microorganisms in the occurrence and development of cardiovascular diseases has been gradually recognized and widely studied. A large number of research data have confirmed that the richness and diversity of intestinal flora in patients with hypertension are decreased compared with healthy people, and intestinal flora is involved in regulating blood pressure through a variety of mechanisms. In the feces of patients with heart failure represented by HFrEF, the diversity of gut microbiota is significantly decreased, and the composition structure of gut microbiota is changed. Pathogenic bacteria such as Campylobacter and Candida are significantly increased, and are related to the severity of the disease, while anti-inflammatory related bacteria such as Blautia are significantly decreased. Gut microbiota can also affect host cardiometabolic processes by regulating metabolites. The distal gut microbiota can promote the production of SCFAs by fermentation processes such as dietary fiber, regulate blood pressure by recognizing specific host receptors, and play an anti-inflammatory role by activating histone acetyltransferase. Gut microbiota in the colon can metabolize unrecycled primary bile acids to produce secondary bile acids, such as deoxycholate, lithocholate, and ursodeoxycholate. Primary bile acids and secondary bile acids directly or indirectly affect cardiovascular function, and regulate atherosclerosis, obesity, metabolism, inflammation, liver pathophysiology by acting on specific receptors. fecal microbiota transplantation (FMT) is the transfer of minimally processed feces from a healthy donor to the gut of a recipient. The purpose is to treat diseases associated with alterations in the gut microbiota, improve the imbalance of gut microbiota, and reestablish a normal functioning gut microbiota. It was previously used for the treatment of recurrent Clostridium difficile infection. In recent years, some countries have classified FMT as tissue transplantation, because feces is not a simple mixture of microorganisms, but a heterogeneous mixture of microorganisms, human cells, water, mucus, and metabolites, which is affected by the donor's own factors (age, lifestyle, etc.). Studies have found that the therapeutic potential of FMT is not limited to gastrointestinal diseases. The loss of gut microbiota alters the composition of the immune system and impairs cardiac repair after MI. The survival and physiological state of mice after fecal reconstitution are improved. Dysbiosis of gut microbiota in metabolic syndrome is associated with a proinflammatory state and impaired mucosal barrier function. Fecal FMT from lean donors improves glucose clearance in obese patients with metabolic syndrome. Fecal microbiota from healthy rats transplanted into hypertensive rats induced by high-salt diet significantly reduced blood pressure in rats, suggesting that FMT is promising for the treatment of patients with chronic hypertension. At present, more and more scholars believe that HFpEF is a metabolic disease. The common comorbidities of HFpEF include obesity, type 2 diabetes, metabolic syndrome, hypertension, coronary atherosclerotic heart disease, and kidney disease, which have been reported to be closely related to intestinal flora in the past. However, the relationship between gut microbiota and HFpEF remains poorly studied. Only a few small sample clinical studies have shown that fecal SCFAs and Trimethylamine N-oxide (TMAO) are altered in HFpEF patients, and TMAO is associated with poor prognosis in HFrEF patients. Subsequently, elevated circulating TMAO in HFpEF patients was found to be positively associated with adverse cardiovascular events such as cardiac death and rehospitalization for heart failure, and these metabolites have been shown to be closely related to gut microbiota. In addition, HFpEF is associated with intestinal epithelial dysfunction, which can easily lead to intestinal congestion or ischemia, change the morphology and permeability of the intestinal wall, and cause changes in the composition and abundance of intestinal flora, suggesting that intestinal flora may play an important regulatory role in HFpEF, a chronic cardiovascular syndrome. Targeting intestinal flora and metabolites is expected to become a new treatment strategy for HFpEF.

This study aims to reveal the role of gut microbiota and metabolites in the regulation of HFpEF and the related mechanisms. Through the establishment of a clinical cohort of HFpEF patients, the changes of gut microbiota and the expression of key metabolites in blood samples of HFpEF patients were confirmed, and their correlation with clinical indicators was analyzed, so as to provide potential biomarkers and therapeutic targets for the diagnosis, prevention and treatment of HFpEF, a major chronic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years old;
2. With symptoms and signs of chronic heart failure, NYHA class II-IV;
3. LVEF≥50% according to the most recent echocardiography before screening, and no previous record of LVEF<50%;
4. BNP >35 pg/mL, or NT-proBNP >125 pg/mL;
5. Comply with at least one of the following:

(1) LVMI ≥ 115g/m2 (men) 95g/m2 (women); (2) RWT > 0.42; R (3) E/e '>15; (4) septal e '<7cm/s or lateral e' <10cm/s or mean e '<8cm/s; (5) TVR>2.8m/s or PASP>35mmHg.

Exclusion Criteria:

Patients with confirmed chronic or acute renal insufficiency (stage II-IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who met the inclusion criteria of this cohort study were consecutively screened in the Department of Cardiovascular Medicine, the First Affiliated Hospital of Nanjing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Death and rehospitalization | 3 years
  All-cause death and rehospitalization due to cardiac causes within 3 years

SECONDARY OUTCOMES:
Health-related quality of life | 3 years.
  Three-year changes in the total score and each component of health-related quality of life (HRQoL) including physical, psychological, and social functioning, all-cause mortality, and cardiogenic rehospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Naning, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kinugasa Y, Nakamura K, Kamitani H, Hirai M, Yanagihara K, Kato M, Yamamoto K. Trimethylamine N-oxide and outcomes in patients hospitalized with acute heart failure and preserved ejection fraction. ESC Heart Fail. 2021 Jun;8(3):2103-2110. doi: 10.1002/ehf2.13290. Epub 2021 Mar 18. PMID 33734604
- [Background] Beale AL, O'Donnell JA, Nakai ME, Nanayakkara S, Vizi D, Carter K, Dean E, Ribeiro RV, Yiallourou S, Carrington MJ, Marques FZ, Kaye DM. The Gut Microbiome of Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2021 Jul 6;10(13):e020654. doi: 10.1161/JAHA.120.020654. Epub 2021 Jul 2. PMID 34212778
- [Background] Wang YC, Koay YC, Pan C, Zhou Z, Tang W, Wilcox J, Li XS, Zagouras A, Marques F, Allayee H, Rey FE, Kaye DM, O'Sullivan JF, Hazen SL, Cao Y, Lusis AJ. Indole-3-Propionic Acid Protects Against Heart Failure With Preserved Ejection Fraction. Circ Res. 2024 Feb 16;134(4):371-389. doi: 10.1161/CIRCRESAHA.123.322381. Epub 2024 Jan 24. PMID 38264909
- [Background] Troseid M, Andersen GO, Broch K, Hov JR. The gut microbiome in coronary artery disease and heart failure: Current knowledge and future directions. EBioMedicine. 2020 Feb;52:102649. doi: 10.1016/j.ebiom.2020.102649. Epub 2020 Feb 12. PMID 32062353
- [Background] Yang T, Richards EM, Pepine CJ, Raizada MK. The gut microbiota and the brain-gut-kidney axis in hypertension and chronic kidney disease. Nat Rev Nephrol. 2018 Jul;14(7):442-456. doi: 10.1038/s41581-018-0018-2. PMID 29760448
- [Background] Sanna S, van Zuydam NR, Mahajan A, Kurilshikov A, Vich Vila A, Vosa U, Mujagic Z, Masclee AAM, Jonkers DMAE, Oosting M, Joosten LAB, Netea MG, Franke L, Zhernakova A, Fu J, Wijmenga C, McCarthy MI. Causal relationships among the gut microbiome, short-chain fatty acids and metabolic diseases. Nat Genet. 2019 Apr;51(4):600-605. doi: 10.1038/s41588-019-0350-x. Epub 2019 Feb 18. PMID 30778224
- [Background] Gomes AC, Hoffmann C, Mota JF. The human gut microbiota: Metabolism and perspective in obesity. Gut Microbes. 2018 Jul 4;9(4):308-325. doi: 10.1080/19490976.2018.1465157. Epub 2018 May 24. PMID 29667480
- [Background] Pinto YM. Heart Failure with Preserved Ejection Fraction - A Metabolic Disease? N Engl J Med. 2023 Sep 21;389(12):1145-1146. doi: 10.1056/NEJMe2309294. Epub 2023 Aug 25. No abstract available. PMID 37622676
- [Background] Luedde M, Winkler T, Heinsen FA, Ruhlemann MC, Spehlmann ME, Bajrovic A, Lieb W, Franke A, Ott SJ, Frey N. Heart failure is associated with depletion of core intestinal microbiota. ESC Heart Fail. 2017 Aug;4(3):282-290. doi: 10.1002/ehf2.12155. Epub 2017 Apr 21. PMID 28772054
- [Background] Pasini E, Aquilani R, Testa C, Baiardi P, Angioletti S, Boschi F, Verri M, Dioguardi F. Pathogenic Gut Flora in Patients With Chronic Heart Failure. JACC Heart Fail. 2016 Mar;4(3):220-7. doi: 10.1016/j.jchf.2015.10.009. Epub 2015 Dec 9. PMID 26682791
- [Background] Hou K, Wu ZX, Chen XY, Wang JQ, Zhang D, Xiao C, Zhu D, Koya JB, Wei L, Li J, Chen ZS. Microbiota in health and diseases. Signal Transduct Target Ther. 2022 Apr 23;7(1):135. doi: 10.1038/s41392-022-00974-4. PMID 35461318
- [Background] Boulange CL, Neves AL, Chilloux J, Nicholson JK, Dumas ME. Impact of the gut microbiota on inflammation, obesity, and metabolic disease. Genome Med. 2016 Apr 20;8(1):42. doi: 10.1186/s13073-016-0303-2. PMID 27098727
- [Background] Steinberg BA, Zhao X, Heidenreich PA, Peterson ED, Bhatt DL, Cannon CP, Hernandez AF, Fonarow GC; Get With the Guidelines Scientific Advisory Committee and Investigators. Trends in patients hospitalized with heart failure and preserved left ventricular ejection fraction: prevalence, therapies, and outcomes. Circulation. 2012 Jul 3;126(1):65-75. doi: 10.1161/CIRCULATIONAHA.111.080770. Epub 2012 May 21. PMID 22615345
- [Background] Pfeffer MA, Shah AM, Borlaug BA. Heart Failure With Preserved Ejection Fraction In Perspective. Circ Res. 2019 May 24;124(11):1598-1617. doi: 10.1161/CIRCRESAHA.119.313572. PMID 31120821
- [Background] Anker SD, Butler J, Filippatos G, Ferreira JP, Bocchi E, Bohm M, Brunner-La Rocca HP, Choi DJ, Chopra V, Chuquiure-Valenzuela E, Giannetti N, Gomez-Mesa JE, Janssens S, Januzzi JL, Gonzalez-Juanatey JR, Merkely B, Nicholls SJ, Perrone SV, Pina IL, Ponikowski P, Senni M, Sim D, Spinar J, Squire I, Taddei S, Tsutsui H, Verma S, Vinereanu D, Zhang J, Carson P, Lam CSP, Marx N, Zeller C, Sattar N, Jamal W, Schnaidt S, Schnee JM, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Preserved Trial Investigators. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. N Engl J Med. 2021 Oct 14;385(16):1451-1461. doi: 10.1056/NEJMoa2107038. Epub 2021 Aug 27. PMID 34449189
- [Background] Solomon SD, McMurray JJV, Claggett B, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Jhund PS, Belohlavek J, Chiang CE, Borleffs CJW, Comin-Colet J, Dobreanu D, Drozdz J, Fang JC, Alcocer-Gamba MA, Al Habeeb W, Han Y, Cabrera Honorio JW, Janssens SP, Katova T, Kitakaze M, Merkely B, O'Meara E, Saraiva JFK, Tereshchenko SN, Thierer J, Vaduganathan M, Vardeny O, Verma S, Pham VN, Wilderang U, Zaozerska N, Bachus E, Lindholm D, Petersson M, Langkilde AM; DELIVER Trial Committees and Investigators. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. N Engl J Med. 2022 Sep 22;387(12):1089-1098. doi: 10.1056/NEJMoa2206286. Epub 2022 Aug 27. PMID 36027570
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2023 Oct 1;44(37):3627-3639. doi: 10.1093/eurheartj/ehad195. No abstract available. PMID 37622666
- [Background] Shah KS, Xu H, Matsouaka RA, Bhatt DL, Heidenreich PA, Hernandez AF, Devore AD, Yancy CW, Fonarow GC. Heart Failure With Preserved, Borderline, and Reduced Ejection Fraction: 5-Year Outcomes. J Am Coll Cardiol. 2017 Nov 14;70(20):2476-2486. doi: 10.1016/j.jacc.2017.08.074. Epub 2017 Nov 12. PMID 29141781
- [Background] Redfield MM, Borlaug BA. Heart Failure With Preserved Ejection Fraction: A Review. JAMA. 2023 Mar 14;329(10):827-838. doi: 10.1001/jama.2023.2020. PMID 36917048
- [Background] Dunlay SM, Roger VL, Redfield MM. Epidemiology of heart failure with preserved ejection fraction. Nat Rev Cardiol. 2017 Oct;14(10):591-602. doi: 10.1038/nrcardio.2017.65. Epub 2017 May 11. PMID 28492288